CLINICAL TRIAL: NCT01120509
Title: Crux Biomedical Evaluation of the Crux Inferior Vena Cava Filter System 2
Brief Title: Crux Biomedical Vena Cava Filter Study - United States
Acronym: RETRIEVE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crux Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Crux02
Record Dates: First submitted 2010-04-29; First posted 2010-05-11 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2012-08

CONDITIONS: Pulmonary Embolism
Keywords: Vena Cava; Vena Cava Filter; Pulmonary Embolism; Venous Thromboembolism; Risk of Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism | interventions — Vena Cava Filters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Crux Vena Cava Filter System (Experimental): Subjects at risk for Pulmonary Embolism
  Interventions: Device: Inferior Vena Cava Filter

INTERVENTIONS:
Device: Inferior Vena Cava Filter — Inplant of filter in inferior vena cava.

SUMMARY:
The purpose of this study is to determine if the Crux Vena Cava Filter System is safe and effective in preventing pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a permanent or temporary risk of Pulmonary Embolism
* Patient or legal guardian must provide written informed consent
* At least one of the following conditions

  * Proven PE
  * Recurrent PE despite adequate anticoagulation
  * Contraindication to anticoagulation
  * Inability to achieve/maintain therapeutic anticoagulation
  * Iliocaval DVT
  * Large, free-floating proximal DVT
  * Massive PE treated with thrombolysis/thrombectomy
  * Chronic PE treated with thrombectomy
  * Procetion during thrombolysis for iliocaval DVT
  * PE with limited cardiopulmonary reserve
  * Poor compliance with anticoagulation medication
  * High risk of injury worsend by anticoagulation
  * Multi-trauma patient with high risk of PE
  * Surgical patients at high risk of PE
  * Medical condition with high risk of PE
* Patient has documented vena cava diameter of 17-28mm
* Patient has IVC anatomy suitable for infra-renal placement
* Patient willing to be available for the appropriate follow up.

Exclusion Criteria:

* Age <18 years old
* Patient has any one of the following conditions

  * Renal vein thrombosis
  * IVC thrombosis extending to te renal veins
  * Duplicate IVC
  * Gonadal vein thrombosis
  * Requires supra-renal placement
* Uncontrolled infectious disease
* Risk of aseptic PE
* Uncontrolled coagulopathy
* Existing inferior vena cava filter implant
* Life expectancy less than 6 months
* Pregnant or planning a pregnancy in the next 6 months
* Condition that inhibits radiographic visualization of the IVC
* Known allergy or intolerance to polytetrafluoroethylene (PTFE) or Nitinol
* Known hypersensitivity to contract which cannot be pretreated
* Access vessels preclude safe insertion of delivery system
* Participation in another drug or device trial
* Unable or unwilling to cooperate with study procedures or required follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 6 Months
  Clinical Success is a composite endpoint consisting of technical success with freedom from pulmonary embolism, filter migration and device related events requiring intervention.

SECONDARY OUTCOMES:
Retrieval Success | 6 Months
Filter Migration | 6 Months
VCF Thrombus | 6 Months
Device Integrity | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mendes, MD, Principal Investigator — University Hospital, Augusta, Georgia, USA
Locations (17):
- United States (17):
  - St. Joseph's Hospital, Orange, California
  - University of California at Irvine Medical Center, Orange, California
  - Univeristy of California at Davis Medical Center, Sacramento, California
  - Christiana Care, Newark, Delaware
  - University of Florida Medical Center, Gainesville, Florida
  - Atlanta Medical Center, Atlanta, Georgia
  - University Hospital, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - St. Francis Hospital, Peoria, Illinois
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Albany Medical Center, Albany, New York
  - Upstate Medical Center, Syracuse, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Jobst Vascular Institute, Toledo, Ohio
  - Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia Medical Center, Charlottesville, Virginia

REFERENCES:
- See also: Smouse H, Mendes R, Bosiers M et al. The RETRIEVE Trial: Safety and Effectiveness of the Retrieval Crux Vena Cava Filter. JVIR 2013; 24:609-621. — http://www.ncbi.nlm.nih.gov/pubmed/23622035